CLINICAL TRIAL: NCT05150964
Title: Measuring Comfort and Clarity Using Low Gain Feature in Pediatric Hearing Aid Users
Brief Title: Measuring Comfort and Clarity With Low Gain Feature in Pediatric Hearing Aid Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SRF-379
Record Dates: First submitted 2021-09-28; First posted 2021-12-09 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental (Experimental): One group will be fit with commercially available hearing aids that will have different program settings
  Interventions: Device: Phonak Audeo hearing aid

INTERVENTIONS:
Device: Phonak Audeo hearing aid — receiver in the canal devices with custom earmolds

SUMMARY:
Comfort and clarity of speech will be measured in hearing impaired children age 8-17 using standard speech processing algorithm with a soft speech enhancer feature, referred to as the Adaptive Situational Gain (ASG) feature in study documents.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of mild, moderate, or moderate-severe sensorineural hearing loss
* Must use oral mode of communication
* must speak English

Exclusion Criteria:

-

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: One group will be fit with commercially available hearing aids that will have different program settings. Each participant will be tested with the study hearing devices in the following conditions:
  1. Hearing device programmed with the NAL (National Acoustic Laboratory) fitting prescription and with the ASG feature both on and off.
  2. Hearing device programmed with the DSL (Desired Sensation Level) fitting prescription and with the ASG feature both on and off.
  For certain speech tests the above conditions will apply but will include testing levels at both a louder level and a softer level.
  Phonak Audeo hearing aid: receiver in the canal devices with non-custom earmolds
Period: Overall Study
Arm/Group | Experimental
Started | 16
Completed | 14
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Experimental: One group will be fit with commercially available hearing aids that will have different program settings
  Phonak Audeo hearing aid: receiver in the canal devices with non-custom earmolds
Arm/Group | Experimental
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 13.7 [9 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Speech Reception Threshold
Description: A familiar spondee word list is presented at varying dB (decibel) levels. Threshold is defined as the lowest dB level at which a correct response occurs for two out of three ascending trials. Testing was completed in two, two-hour test sessions occurring two weeks apart. A different fitting prescription, NAL (National Acoustic Laboratory) or DSL (Desired Sensation Level) was selected for each test session, and counterbalanced across participants. Each session consisted of testing with the ASG (Adaptive Situational Gain) feature on and off. The lower the number (dB level), the softer the participant is able to repeat the words correctly two out of three times.
Time Frame: Initial appointment (day 1 of study) and 2nd appointment (Day 14 of study)
Population: Participants who were fit with study hearing aids and completed at least one two-hour test session.
Measure: Mean (Standard Deviation); unit: dB HL (decibels hearing level)
Groups:
- Experimental: One group will be fit with commercially available hearing aids that will have different program settings. Each participant will be tested with the study hearing devices in the following conditions:
  1. Hearing device programmed with the NAL (National Acoustic Laboratory) fitting prescription and with the ASG feature both on and off.
  2. Hearing device programmed with the DSL (Desired Sensation Level) fitting prescription and with the ASG feature both on and off.
  Phonak Audeo hearing aid: receiver in the canal devices with non-custom earmolds
Arm/Group | Experimental
Number analyzed (Participants) | 15
dB HL (decibels hearing level)
  NAL Fitting with ASG Off | 27 (8)
  NAL Fitting with ASG ON | 27 (7)
  DSL Fitting with ASG Off | 24 (8)
  DSL Fitting with ASG On | 24 (6)
Statistical Analysis 1: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (NAL/National Acoustic Laboratory or DSL/Desired Sensation Level) and ASG (Adaptive Situational Gain) setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. Null hypothesis: The hearing aid fitting prescription will have no effect on the speech reception thresholds; Test type: Other; p < 0.05, Mixed Models Analysis — Significance was indicated by p <. 05, Cohen's d was calculated to indicate effect size
Statistical Analysis 2: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (NAL/National Acoustic Laboratory or DSL/Desired Sensation Level) and ASG (Adaptive Situational Gain) setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. Null hypothesis: The ASG setting will have no effect on the speech reception threshold; Test type: Other; p > 0.05, Mixed Models Analysis — Significance was indicated by p <. 05, Cohen's d was calculated to indicate effect size

2. Primary Outcome: Word Recognition Score With Words Presented at 40 dB SPL (Decibel Sound Pressure Level) and 70 dB SPL.
Description: Familiar monosyllabic word list presented at 40 dB and 70 dB. Percentage of words correctly repeated is calculated. Testing was completed in two, two-hour test sessions occurring two weeks apart. A different fitting prescription, NAL (National Acoustic Laboratory) or DSL (Desired Sensation Level) was selected for each test session and counterbalanced across participants such that one test session consisted of testing with one prescription, either NAL or DSL, but with both levels (40 and 70 dB) and with both ASG (Adaptive Situational Gain) settings, on and off. The higher the score, the better the word recognition in each condition.
Time Frame: Initial appointment (Day 1 of study) and 2nd appointment (day 14 of study)
Population: Participants who were fit with study hearing aids and completed at least one two-hour test session.
Measure: Mean (Standard Deviation); unit: percentage of words correctly repeated
Groups:
- Experimental: One group will be fit with commercially available hearing aids that will have different program settings. Each participant will be tested with the study hearing devices in the following conditions:
  1. Hearing device programmed with the NAL (National Acoustic Laboratory) fitting prescription and with the ASG feature both on and off, and stimuli presented at both 40 dB and 70 dB.
  2. Hearing device programmed with the DSL (Desired Sensation Level) fitting prescription and with the ASG feature both on and off, and stimuli presented at both 40 dB and 70 dB.
  For certain speech tests the above conditions will apply but will include testing levels at both a louder level and a softer level.
  Phonak Audeo hearing aid: receiver in the canal devices with non-custom earmolds
Arm/Group | Experimental
Number analyzed (Participants) | 15
percentage of words correctly repeated
  % correct at 40 dB, NAL fitting, ASG Off | 52 (24)
  % correct at 40 dB, NAL fitting, ASG On | 63 (26)
  % correct at 40 dB, DSL fitting, ASG Off | 69 (21)
  % correct at 40 dB, DSL fitting, ASG On | 75 (22)
  % correct at 70 dB, NAL fitting, ASG Off | 92 (10)
  % correct at 70 dB, NAL fitting, ASG On | 95 (5)
  % correct at 70 dB, DSL fitting, ASG Off | 95 (6)
  % correct, DSL fitting, ASG On | 96 (7)
Statistical Analysis 1: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null Hypothesis: The ASG setting will have no effect on the Word Recognition Scores; Test type: Other; p < 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size
Statistical Analysis 2: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null Hypothesis: The presentation level will have no effect on the Word Recognition Scores; Test type: Other; p < 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size
Statistical Analysis 3: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null Hypothesis: Hearing aid prescription will have no effect on the Word Recognition Scores; Test type: Other; p < 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size

3. Primary Outcome: Multi-word Recognition at 40 dB SPL and 70 dB SPL
Description: Out of a list of seven words, the participant repeats back as many words as they can recall. Percentage of correct words repeated back is calculated. Testing was completed in two, two-hour test sessions occurring two weeks apart. One fitting prescription, NAL (National Acoustic Laboratory) or DSL (Desired Sensation Level) was selected for each test session and counterbalanced across participants such that one test session consisted of testing with one prescription, either NAL or DSL, but with both levels (40 and 70 dB) and with both ASG (Adaptive Situational Gain) settings, on and off. A higher percentage score indicates better multi-word recognition.
Time Frame: Initial appointment (Day 1 of study) and 2nd appointment (Day 14 of study)
Population: Participants who were fit with study hearing aids and completed at least one two-hour test session.
Measure: Mean (Standard Deviation); unit: percentage of words correctly repeated
Arm/Group | Experimental
Number analyzed (Participants) | 15
percentage of words correctly repeated
  % correct at 40 dB for NAL fitting, ASG Off | 48 (20)
  % correct at 40 dB for NAL fitting, ASG On | 56 (16)
  % correct at 40 dB for DSL fitting, ASG Off | 51 (16)
  % correct at 40 dB for DSL fitting, ASG On | 54 (16)
  % correct at 70 dB, NAL fitting, ASG Off | 66 (17)
  % correct at 70 dB, NAL fitting, ASG On | 67 (13)
  % correct at 70 dB, DSL fitting, ASG Off | 63 (13)
  % correct at 70 dB, DSL fitting, ASG On | 67 (13)
Statistical Analysis 1: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null hypothesis: Presentation level will have no effect on multi-word recognition scores; Test type: Other; p < 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size
Statistical Analysis 2: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null hypothesis: The ASG setting will have no effect on multi-word recognition scores; Test type: Other; p > 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size
Statistical Analysis 3: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null hypothesis: Hearing aid prescription will have no effect on multi-word recognition scores; Test type: Other; p > 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size

4. Primary Outcome: Nonword Detection Presented at 40 dB SPL and at 70 dB SPL.
Description: A list of 10 3-word phrases are presented to the participant. The participant indicates if the phrase contains a nonsense word by selecting the numbered response button (i.e. "1", "2", or "3") that corresponds to the position oof the nonsense word in the phrase. Testing was completed in two, two-hour test sessions occurring two weeks apart. A different fitting prescription, NAL (National Acoustic Laboratory) or DSL (Desired Sensation Level) was selected for each test session and counterbalanced across participants such that one test session consisted of testing with one prescription, either NAL or DSL, but with both levels (40 and 70 dB) and with both ASG (Adaptive Situational Gain) settings, on and off. . The score is the percent correct, a higher score is better.
Time Frame: Initial appointment (Day 1 of study) and 2nd appointment (day 14 of study)
Population: Participants who were fit with study hearing aids and completed at least one two-hour test session.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Experimental
Number analyzed (Participants) | 15
percentage of correct responses
  % correct at 40 dB, NAL fitting formula, ASG Off | 65 (15)
  % correct at 40 dB, NAL fitting with ASG On | 68 (13)
  % correct at 40 dB, DSL fitting, ASG Off | 73 (18)
  % correct at 40 dB, DSL fitting, ASG On | 71 (12)
  % correct at 70 dB, NAL fitting, ASG Off | 89 (7)
  % correct at 70 dB, NAL fitting, ASG On | 87 (7)
  % correct at 70 dB, DSL fitting, ASG Off | 88 (9)
  % correct at 70 dB, DSL fitting, ASG On | 87 (7)
Statistical Analysis 1: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null hypothesis: Presentation level will have no effect on Nonword Detection scores; Test type: Other; p < 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size
Statistical Analysis 2: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null hypothesis: Hearing aid prescription will have no effect on Nonword Detection scores; Test type: Other; p < 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size
Statistical Analysis 3: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null hypothesis: The ASG setting will have no effect on Nonword Detection scores; Test type: Other; p > 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size

5. Primary Outcome: Rapid Word Learning With Stimuli Presented at 40 dB SPL and at 70 dB SPL.
Description: A word learning task used to determine participant's ability to associate novel/nonsense words with novel images as rapidly as possible. Five nonsense words are paired with five novel images displayed on response buttons. The words are presented randomly 10 times each. The participant selects one picture per word. Scores are presented as percent correct. A higher percentage indicates better word learning. Testing was completed in two, two-hour test sessions occurring two weeks apart. A different prescription, NAL (National Acoustic Laboratory) or DSL (Desired Sensation Level) was selected for each test session and counterbalanced across participants such that one test session consisted of testing with one prescription, either NAL or DSL, but with both levels (40 and 70 dB) and with both ASG (Adaptive Situational Gain) settings, on and off.
Time Frame: Initial appointment (Day 1 of study) and 2nd appointment (day 14 of study)
Population: Participants who were fit with study hearing aids and completed at least one two-hour test session.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Experimental
Number analyzed (Participants) | 15
percentage of correct responses
  % correct at 40 dB, NAL fitting, ASG Off | 68 (23)
  % correct at 40 dB, NAL fitting, ASG On | 76 (18)
  % correct at 40 dB, DSL fitting, ASG Off | 70 (22)
  % correct at 40 dB, DSL fitting, ASG On | 73 (20)
  % correct at 70 dB, NAL fitting, ASG Off | 69 (18)
  % correct at 70 dB, NAL fitting, ASG On | 73 (16)
  % correct at 70 dB, DSL fitting, ASG Off | 67 (20)
  % correct at 70 dB, DSL fitting, ASG On | 70 (21)
Statistical Analysis 1: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null hypothesis: The ASG setting will have no effect on Rapid Word Learning scores; Test type: Other; p > 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size
Statistical Analysis 2: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null hypothesis: Presentation level will have no effect on Rapid Word Learning scores; Test type: Other; p > 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size
Statistical Analysis 3: Comparison: Experimental; A Linear Mixed Model Analysis was performed. The hearing aid prescription (DSL, NAL) and ASG setting (on, off) were entered as fixed factors while the individual participants were entered as a random factor. An additional fixed factor of presentation level (40, 70 dB SPL) was added to the analyses. Null hypothesis: Hearing aid prescripton will have no effect on Rapid Word Learning scores; Test type: Other; p > 0.05, Mixed Models Analysis — Significance was indicated by p <. 05 and Cohen's d was calculated to indicate effect size

6. Primary Outcome: Subjective Preference for the Adaptive Situational Gain Feature With Each Fitting Formula
Description: Participants will rank preference for the ASG feature (either on or off) in each fitting (NAL and DSL) after listening to audio file.
Time Frame: 2nd appointment (day 14 of study)
Population: Participants who were fit with study hearing aids and completed both two-hour test sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 14
Participants
  Number of participants preferring ASG Off with NAL fitting | 2
  Number of participants preferring ASG On with NAL fitting | 2
  Number of participants preferring ASG Off with DSL fitting | 7
  Number of participants preferring ASG On with DSL fitting | 3

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT05150964/Prot_SAP_000.pdf